CLINICAL TRIAL: NCT01685866
Title: Difficult Venous Access in Pediatric Anesthesia: Evaluation of a New Medical Device in Multicenter Trial.
Brief Title: 3V- Improve Venous Access in Pediatric Anesthesia
Acronym: 3V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SC/DM_JDS_2012-1_V1.0-20120605
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Cardiovascular Diseases
Keywords: anesthesia; venous access
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vein-Viewer Vision (Other): A medical device called Vein-Viewer Vision
  Interventions: Device: Vein-Viewer Vision
- no medical device (No Intervention): in the second arm, we use no medical device

INTERVENTIONS:
Device: Vein-Viewer Vision — A medical device called Vein-Viewer Vision
  Arms: Vein-Viewer Vision

SUMMARY:
Our hypothesis is that a new medical device called Vein-Viewer Vision helps to see peripheral veins in children having forecasted difficult venous access and could facilitate the venous access.The main goal is to reduce the time necessary to get a venous access during the inhalation anesthesia induction.

DETAILED DESCRIPTION:
Randomized study comparing the delay of peripheral access with or without using the device. Monosite study, including children undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* children aged less than 7
* DIVA score ≥ 4
* patient needing venous peripheral access for general anesthesia

Exclusion Criteria:

* no social security
* opposition of the parent(s) to the participation of their child in the trial

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 311 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
reduce the time necessary to find the venous access during inhalation anesthesia induction | 1 day of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Devys, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (2):
- France (2):
  - Fondation ophtalmologique Adolphe de Rothschild, Paris, Île-de-France Region
  - Robert Debré Hospital, APHP, Paris, Île-de-France Region

REFERENCES:
- [Derived] Gras S, Roy-Gash F, Bruneau B, Salvi N, Colas AE, Skhiri A, Orliaguet G, Dahmani S, Devys JM. Reducing the time to successful intravenous cannulation in anaesthetised children with poor vein visibility using a near-infrared device: A randomised multicentre trial. Eur J Anaesthesiol. 2021 Aug 1;38(8):888-894. doi: 10.1097/EJA.0000000000001467. PMID 33606421